CLINICAL TRIAL: NCT01832012
Title: Practical Skill Retention in Medical Students: Improving Cardiopulmonary Resuscitation With Hands-On Practice
Brief Title: Basic Life Support Cardiopulmonary Resuscitation Refresher in MS2 at St George's University
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Windward Islands Research and Education Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: SGUCPR1
Record Dates: First submitted 2013-04-09; First posted 2013-04-15 (Estimated); Last update posted 2013-04-15 (Estimated); Status verified 2013-04

CONDITIONS: Cardiopulmonary Resuscitation Skill Retention in Medical Students
Keywords: Eliciting which type of refresher provides the greatest improvement in BLS CPR skills.
MeSH Terms: interventions — Multimedia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Video refresher (Active Comparator): Group 3, received 7 minute video refresher prior to examination.
  Interventions: Other: Multimedia
- Video refresher and hands-on practice (Experimental): Group 4, received same 7 minute video refresher, along with hands-on practice along with the video on a Laerdal BLS manikin.
  Interventions: Other: Multimedia; Other: Hands-on practice
- No intervention (No Intervention): Group 2

INTERVENTIONS:
Other: Multimedia — AHA specific BLS refresher video, 7 minutes in length.
  Arms: Video refresher; Video refresher and hands-on practice
Other: Hands-on practice — Hands-on BLS CPR practice on a Laerdal BLS manikin.
  Arms: Video refresher and hands-on practice

SUMMARY:
175 second year medical students were assessed on their BLS CPR skill retention after an approximate one year after taking the initial certification class, and the investigators assessed which type of refresher course would be most effective in improving the students' CPR skills. Group 2 had no refresher, Group 3 had a multimedia refresher, and Group 4 had the same multimedia refresher plus hands on practice on a Laerdal BLS manikin. The investigators hypothesized that Group 4 would perform CPR skills with the highest competency compared to the other two groups.

ELIGIBILITY:
Inclusion Criteria:

* Voluntary second year medical student

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 175 (Actual)
Dates: Start 2012-07; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Chest compressions | 1 session
  Chest compressions were measured on a Laerdal Resusci-Anne recording manikin for each subject.
Bag Valve Mask ventilations | 1 session
  Bag Valve Mask ventilations were measured for each subject on a Laerdal Resusci-Anne recording manikin.

CONTACTS AND LOCATIONS:
Overall Officials: Alexander M Dabrowiecki, BS, Principal Investigator — St. George's University
Locations (1):
- St. George's University, True Blue, Saint George's, Grenada